CLINICAL TRIAL: NCT03444974
Title: Addiction and Substance Dependence in Adolescence - Neurobiological Pathomechanisms and Treatment Evaluation
Brief Title: Addiction in Adolescence - Pathomechanisms and Treatment Evaluation
Acronym: MATRIX-A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MATRIX-A
Record Dates: First submitted 2018-02-06; First posted 2018-02-26 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Substance Use Disorders; Adolescent Behavior
Keywords: drugs; youth; adolescence; abuse; dependence; Tetrahydrocannabinol (THC); Methamphetamine (Crystal Meth); Marihuana; comorbidity; treatment; etiopathology; sociodemographics; Saxony; MATRIX; Psychotherapy
MeSH Terms: conditions — Substance-Related Disorders; Adolescent Behavior; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: Symptom reduction in the treatment group (adolescent patients with substance abuse and dependency) in comparison to age and gender matched waiting-list and healthy controls. Changes in parental stress levels and parenting skills in the treatment group parents in comparison to waiting-list parents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Patient therapy group (Active Comparator): * Adolescents with substance use disorders
  * Receiving an adapted treatment according to the MATRIX-A therapy
  Interventions: Other: adapted treatment according to the MATRIX-A therapy
- Parental therapy group (Active Comparator): * Parents of adolescents with substance use disorders
  * Receiving an adapted treatment according to the MATRIX-A therapy
  Interventions: Other: adapted treatment according to the MATRIX-A therapy
- Patient waiting list group (No Intervention): * Adolescents with substance use disorders
  * On the waiting list for receiving a MATRIX-A therapy
- Parental waiting list group (No Intervention): * Parents of adolescents with substance use disorders
  * On the waiting list for receiving a MATRIX-A therapy
- control group (No Intervention): * Adolescents with no history of substance use disorders
  * no other intake of psychotropic substances such as psychotropic medication

INTERVENTIONS:
Other: adapted treatment according to the MATRIX-A therapy — cognitive and behavioral treatment of drug abuse/dependency issues, as well as connected parameters
  Arms: Parental therapy group; Patient therapy group

SUMMARY:
This study aims to investigate the sociodemographic background as well as psychiatric comorbidities of adolescent substance users with substance use disorders. The study simultaneously evaluates biomarkers of stress and addiction, including long-term cortisol levels from hair samples and gene methylation in blood samples associated with substance use.

Our study also adapts, rolls out, and evaluates an evaluated multimodal treatment manual wich was originally intended for stimulant drug users (MATRIX). We adopt this manual to the needs and specifics of adolescents (MATRIX-A, A=adolescents) with substance use disorders of any substance, including cannabis, methamphetamine, and alcohol. Adolescents will receive group therapy sessions, individual therapy sessions, and medication if needed, while parents or professional caretaker will receive group sessions. Therapy outcomes will be examined in addition to parental distress and parenting skills.

DETAILED DESCRIPTION:
As numbers of adolescent drug abuse have grown rapidly within the last couple of years, research on youth drug abuse and dependency has taken a new and vital role within the public healthcare system. For this reason, it is crucial to find new ways to effectively integrate adolescent patients into the health care system, as well as assign them to treatment options tailor made for the specific challenges and needs of this population. This study aims to investigate (a) sociodemographic background and psychiatric comorbidities in connection with adolescent substance abuse and dependence to enhance understanding of epidemiologic risk factors for developing drug dependency in adolescence, as well as benefit future treatment options.

It further aims to investigate (b) molecular and epigenetic mechanisms of addiction disorders in adolescents by analyzing methylation pattern, as well as proteome analysis of peripheral immune markers. The investigator's aim is a better understanding of the multimodal biological underpinnings of risk/resilience for addiction in youth on the molecular, cellular and circuit levels with a special focus on the changes within the stress and immune system in patients with addiction disorders and their family members.

Another research interest of this study concerns (c) adapting and evaluating new treatment options, tailor made for the adolescent population. For this reason the investigators aim to adapt, implement and evaluate a therapeutic program according to the MATRIX manual for the treatment of substance abuse, which consists of two group therapies for patients, as well as their parents (Evaluation time points: T0, T1, and T2).

Last, this study aims to (d) evaluate parental stress levels, parental communication skills and knowledge in connection with adolescent substance abuse.

ELIGIBILITY:
Adolescents:

Inclusion Criteria:

* Age 12.00-17.99
* Therapy / wait list group: current substance use disorder
* Controls: no history of substance use disorders

Exclusion Criteria:

* Preexisting neurological diseases
* Diseases of or with involvement of the central nervous system
* Intelligence quotient (IQ) < 70
* Diseases concerning the adrenal gland, pituitary gland or hypothalamus
* Acute viral diseases during T0, T1, T2
* Controls:

  * Drug intake modulating the central nervous system
  * Main psychiatric disorders
  * Current substance use

Parents:

Inclusion Criteria:

* At least one child/protégé with problematic substance abuse
* No current substance abuse on their own
* At least one parent must be eligible to participate in the group

Exclusion Criteria:

* Current substance abuse

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Sociodemographic background | T0
  Sociodemographic background of adolescents with substance use disorders via self-constructed items:
  * age (in years)
  * gender (male/female)
  * highest education (primary school/ currently in high school/ dropped out of school/ finished compulsory school/ finished apprenticeship/ currently doing apprenticeship)
  * migration background (no/ yes > asks for specification)
  * nationality (German/ other > asks for specification)
  * relationship status (single/ married/ separated/ divorced/ widowed/ civil union/ domestic partnership/ other > asks for specification)
Aim 2: Psychiatric comorbidities - MINI-KID | T0, T1, T2
  Current psychiatric comorbidities according to Diagnostic and Statistic Manual of Mental Disorders, 5th Ed. (DSM-5) assessed via Mini International Neuropsychiatric Interview for Children and Adolescents (MINI KID), a structured diagnostic interview. Single interview questions rated (yes / no). DSM-5 diagnoses for past month (or other if specified) in accordance with MINI-KID scoring algorithms.
Aim 2: Change in substance use | T0, T1, T2
  Changes in self-reported substance use between T0, T1, T2. Assessed via quantity and frequency questions for different substance categories.
Aim 3: Changes in biomarkers related to substance use disorders | T0, T1, T2
  * cumulative stress: hair cortisol levels in a single hair sample. Measured in ng/ml.
  * epigenetic changes: methylation pattern in a single blood sample. Measured in %.
  * immunological changes: immune marker Interleukin-6 in a single blood sample. Measured in ng/ml.
Aim 4: Subjective therapy outcomes | T0, T1, T2
  * Evaluation of possible therapy effects (e.g. knowledge, relapse prevention skills, emotions/affects, maintenance self-efficacy, motivation, stress tolerance) with 5-point Likert options (not at T0).
  * Substance use disorder severity assessed via Drug Use Disorders Identification Test (DUDIT). Measured in a test persons's scoring number on the DUDIT scale. Change from baseline DUDIT score to T1 and T2 DUDIT scores.
Aim 4: Objective therapy outcomes | between T0 and T1
  - objective: Abstinence / relapse based on random drug urine tests for illicit substance use during therapy sessions.
Aim 5: Change in baseline parenting skills | T0, T1
  Assessment of parenting skills (communication skills) via descriptive self-reports. Change from T0 to T1. Measured in self-reported description of change.
Aim 5: Change in baseline parental stress reports - ESF | T0, T1, T2
  Change from self-reported baseline parent stress level to T1 anjd T2 parental stress levels. Assessed via a German questionnaire assessing the amount of parental stress (ESF). Stress factors within everyday parent life are being measured with help of 38 items, which are being scored on a 4-point scale that ranges from 0(disagree) to 3 (completely agree). All items can be assigned to 4 different areas of stress, being social support (7 items, total score 0-21 points), workload and restrictions (7 items, total score 0-21 points), social support (7 items, total score 0-21 points) and cooperative partnership (7 items, total score 0-21). High scores report high stress levels.

SECONDARY OUTCOMES:
Emotional, behavioral and social problems of adolescents - Self-Rating (YSR) | Baseline data collection
  Emotional, behavioral and social problems associated with adolescents with substance use disorders: Data collection of existence of emotional/behavioral/social problems with help of the Youth Self-Report (YSR). Measured in a person's scoring on 8 different scales (anxious/depressed, withdrawn/depressed, somatic complaints, social problems, thought problems, attention problems, rule-breaking behavior, aggressive behavior) as well as a total score.
Emotional, behavioral and social problems of adolescents - Parental Rating (CBCL) | T0, T1, T2
  Emotional, behavioral and social problems associated with adolescents with substance use disorders: Data collection of existence of emotional/behavioral/social problems with help of the Child Behavior Checklist (CBCL). Measured in a person's scoring on 8 different scales (anxious/depressed, withdrawn/depressed, somatic complaints, social problems, thought problems, attention problems, rule-breaking behavior, aggressive behavior) as well as a total score.
Adolescent depressivity - BDI-II | T0, T1, T2
  Psychiatric comorbidities associated with adolescents with substance use disorders: Data collection with help of the Beck Depression Inventory (BDI-II). Measured in a test persons's scoring number on the scale.
Mental distress - Brief Symptom Checklist | T0, T1, T2
  Psychiatric comorbidities associated with adolescents with substance use disorders: Data collection with help of the Brief Symptom Checklist (BSCL). Current amount of mental distress is measured in a person's numerical global severity index.
Adolescent satisfaction with life | T0, T1, T2
  Psychiatric comorbidities associated with adolescents with substance use disorders: Data collection with help of the Satisfaction With Life Scale (SWLS). The scale is designed to measure global cognitive judgments of one's life satisfaction with help of 5 items using a 7-point scale that ranges from 7 strongly agree to 1 strongly disagree. Scoring benchmarks: extremely dissatisfied (5-9), dissatisfied (10-14), slightly dissatisfied (15-19), neutral (20), slightly satisfied (21-25), satisfied (26-30), extremely satisfied (31-35).

CONTACTS AND LOCATIONS:
Overall Officials: Veit Roessner, Prof. Dr., Study Director — Technische Universität Dresden, Universitätsklinikum C.G.C. Dresden
Locations (1):
- Department of Child and Adolescent Psychiatry and Psychotherapy, University Hospital C.G.Carus, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zweben JE, Cohen JB, Christian D, Galloway GP, Salinardi M, Parent D, Iguchi M; Methamphetamine Treatment Project. Psychiatric symptoms in methamphetamine users. Am J Addict. 2004 Mar-Apr;13(2):181-90. doi: 10.1080/10550490490436055. PMID 15204668
- [Background] Warden D, Sanchez K, Greer T, Carmody T, Walker R, Dela Cruz A, Toups M, Rethorst C, Trivedi MH. Demographic and clinical characteristics of current comorbid psychiatric disorders in a randomized clinical trial for adults with stimulant use disorders. Psychiatry Res. 2016 Dec 30;246:136-141. doi: 10.1016/j.psychres.2016.09.007. Epub 2016 Sep 15. PMID 27693866
- [Background] Rawson RA, Marinelli-Casey P, Anglin MD, Dickow A, Frazier Y, Gallagher C, Galloway GP, Herrell J, Huber A, McCann MJ, Obert J, Pennell S, Reiber C, Vandersloot D, Zweben J; Methamphetamine Treatment Project Corporate Authors. A multi-site comparison of psychosocial approaches for the treatment of methamphetamine dependence. Addiction. 2004 Jun;99(6):708-17. doi: 10.1111/j.1360-0443.2004.00707.x. PMID 15139869
- [Derived] Basedow LA, Kuitunen-Paul S, Wiedmann MF, Roessner V, Golub Y. Evaluation of the multimodal DELTA therapy for adolescents with substance use disorders: an exploratory pilot trial. Front Psychiatry. 2024 Jan 3;14:1284342. doi: 10.3389/fpsyt.2023.1284342. eCollection 2023. PMID 38234368